CLINICAL TRIAL: NCT00809250
Title: Vaccination With Lethally Irradiated Autologous Myeloblasts With Granulocyte Macrophage-colony Stimulating Factor Secreting K562 Cells (GM-K562) in Patients With Advanced MDS or AML After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Vaccination With GM-K562 Cells in Patients With Advanced Myelodysplastic Syndrome (MDS) or Acute Myeloid Leukemia (AML) After Allogeneic Hematopoetic Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Vincent T. Ho, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-160
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Acute Myeloid Leukemia; Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome-Refractory Anemia With Excess Blasts
Keywords: vaccination; AML; CMML; MDS-RAEB
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GM-K562/leukemia cell vaccine (Experimental): Biological/Vaccine: GM-K562/leukemia cell vaccine Cultured cell line genetically changed to secrete GM-CSF mixed with irradiated leukemia cells obtained from the participant. A total of 6 vaccine will be given. Vaccines 1-3 will be given once a week. Vaccines 4-6 will be given every other week.
  Interventions: Biological: GM-K562/leukemia cell vaccine

INTERVENTIONS:
Biological: GM-K562/leukemia cell vaccine — Cultured cell line genetically changed to secrete GM-CSF mixed with irradiated leukemia cells obtained from the participant. A total of 6 vaccine will be given. Vaccines 1-3 will be given once a week. Vaccines 4-6 will be given every other week.

SUMMARY:
The purpose of this research study is to determine if the GM-K562/leukemia cell vaccine can be safely given soon after allogeneic marrow or blood stem cell transplant. The GM-K562/leukemia cell vaccine is composed of a cultured cell line that has been genetically modified to secrete GM-CSF, a naturally occuring substance in the body that stimulates the immune system. The vaccine is a mixture of the GM-K562 cells (radiated to prevent them from growing in the participants body) with the participant's previously frozen and killed leukemia cells. By mixing the GM-K562 with the leukemia cells, we would like to study whether this vaccine combination will stimulate the participant's new immune system to recognize and fight against their MDS/AML cancer cells.

DETAILED DESCRIPTION:
* Participants will be given the GM-K562/Leukemia call vaccine as in injection under the skin a total of six times. The first 3 vaccines will be given weekly and vaccines 4 through 6 will be given every other week. Therefore, it is expected that the vaccines will be completed over a period of 9 weeks.
* During the 9 week vaccination period, participants will have physical exams to monitor for any side effects or graft-versus-host disease (GVHD). Bone marrow biopsies will be performed a the time of enrollment for this study, 4 weeks after completion of 6 GM-K562/Leukemia cell vaccines, and 1 year after the participants transplant.
* As a way of testing whether the GM-K562/Leukemia cell vaccine is triggering any immune response to the participants leukemia, we will be injecting a small amount of leukemia cells (after they are killed with radiation) under the participants skin to see if the body will generate a reaction to the leukemia cells. This test is called a leukemia cell delayed hypersensitivity test (DTH). This test will be performed three times during the study, on the weeks of the 1st vaccine, 5th vaccine and 4 weeks after the 6th vaccine.
* There are a total of 5 skin biopsies required as part of this study. Biopsies will be taken from the vaccination sites 2-3 days after the first and fifth vaccine. Similar biopsies will be taken from the DTH sites after the 1st vaccination, 5th vaccination and 4-6 weeks after the 6th vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have received an allogeneic bone marrow or peripheral blood stem cell transplant for AML, meeting one of the following: 1) AML arising from MDS or MDP 2)AML CR1 associated with high risk cytogenetics 3) AML transplanted in induction failure or relapse 4) AML transplanted in second remission or beyond 5) AML in patient 60 years or older
* Patients who have received an allogeneic bone marrow or peripheral blood stem cell transplant for MDS-RAEB or CMML
* 18 years of age or older
* Donor is a related or unrelated donor who is at least 9/10 matched at HLA-A, B, C, DRB1, and DQB1 by antigen level typing at class 1 and allele level typing at class II
* Recipients of myeloablative or reduced intensity conditioning transplants are eligible
* Patient must have sufficient autologous tumor cells banked at DFCI (on companion tissue banking protocol) for vaccine generation prior to transplantation
* No active GVHD requiring systemic corticosteroid therapy
* No conditions requiring systemic corticosteroid therapy greater than or equal to 20mg methylprednisolone or equivalent
* No uncontrolled infection
* Adequate hematopoietic engraftment with ANC >500 off growth factor support, and platelet >10k without transfusion
* No non-hematologic toxicity of CTC Grade 3 or greater
* ECOG Performance Status 0-2

Exclusion Criteria:

* Recipients of cord blood transplant
* Patients with uncontrolled CNS disease
* Patients with relapsed/persistent disease after transplant who are expected to require rapid withdrawal of immune suppression, cytoreductive therapy, or have a life expectancy of < 3 months
* Concurrent participation in other transplant clinical trials where GVHD and/or disease relapse are primary endpoints
* Patients deemed medically or psychologically unfit by treating physician or study investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2008-11 (Actual); Primary Completion 2011-05 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
To assess the safety of vaccination, as measured by vaccine related reactions and incidence of grade III-IV acute GVHD. | 2 years

SECONDARY OUTCOMES:
To assess the efficacy of vaccination with GM-K562/leukemia cell vaccine following allogeneic stem cell transplantation in this patient population. | 2 years
To characterize the biologic responses and leukemia specific immune responses after vaccination with GM-K562/leukemia cell vaccine following allogeneic stem cell transplant. | 2 years
To determine duration of disease response, disease free and overall survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Ho, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States